CLINICAL TRIAL: NCT03125395
Title: A Phase 3, Rollover Study to Evaluate the Safety of Long-term Treatment With Lumacaftor/Ivacaftor Combination Therapy in Subjects Aged 2 Years and Older With Cystic Fibrosis, Homozygous for the F508del-CFTR Mutation
Brief Title: A Rollover Safety Study of Lumacaftor/Ivacaftor in Subjects Aged 2 Years and Older With Cystic Fibrosis, Homozygous for the F508del-CFTR Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX16-809-116; 2019-003112-31 (EudraCT Number)
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Results first posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor, ivacaftor drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LUM/IVA (Experimental): LUM/IVA granules or tablets were administered orally every 12 hours (Participants aged 2 through 5 years received LUM 100 mg/IVA 125 mg granules or LUM 150 mg/IVA 188 mg granules based on body weight. Participants ≥6 years of age were to receive LUM 200 mg/IVA 250 mg tablets). Doses were adjusted upward for changes in weight and age.
  Interventions: Drug: LUM/IVA

INTERVENTIONS:
Drug: LUM/IVA — Participants received LUM/IVA every q12h.
  Other Names: VX-809/VX-770; lumacaftor/ivacaftor

SUMMARY:
A Rollover Safety Study of Lumacaftor/Ivacaftor in Subjects Aged 2 Years and Older With Cystic Fibrosis, Homozygous for F508del.

ELIGIBILITY:
Inclusion Criteria:

Subjects entering the Treatment Cohort must meet the following criteria:

* Completed 24 weeks of LUM/IVA treatment and the Safety Follow-up Visit in Study VX15-809-115 Part B (Study 115B, NCT02797132)
* Willing to remain on a stable CF medication regimen through the Safety Follow-up Visit

Subjects entering the Observational Cohort must meet 1 of the following criteria:

* Completed 24 weeks of LUM/IVA treatment and the Safety Follow-up Visit in Study 115B, but do not want to enroll in the Treatment Cohort.
* Received at least 4 weeks of LUM/IVA treatment and completed visits up to Week 24 and the Safety Follow-up Visit, if required, of Study 115B but are not taking LUM/IVA at the end of the Study 115B Treatment Period (i.e., Week 24) because of a drug interruption and either did not receive Vertex approval to enroll in the Treatment Cohort or do not want to enroll in the Treatment Cohort.
* Permanently discontinued LUM/IVA in Study 115B after receiving at least 4 weeks of treatment and remained in the study from the time of treatment discontinuation through the Week 24 Visit and Safety Follow-up Visit, if required.

Exclusion Criteria (Treatment Cohort Only):

* Prematurely discontinued LUM/IVA treatment in Study 115B.
* History of any comorbidity or laboratory abnormality that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering LUM/IVA to the subject
* History of drug intolerance or other serious reactions to LUM/IVA in Study 115B that would pose an additional risk to the subject in the opinion of investigator, and which should be discussed with the Vertex medical monitor.
* Subjects with a history of allergy or hypersensitivity to LUM/IVA.
* Liver function test (LFT) abnormality meeting criteria for LUM/IVA treatment interruption at the completion of Study 115B, for which no convincing alternative etiology is identified.
* QTc value at the completion of Study 115B that would pose an additional risk to the subject in the opinion of investigator, and which should be discussed with the Vertex medical monitor
* History of poor compliance with LUM/IVA and/or procedures in Study 115B as deemed by the investigator.
* Participation in an investigational drug trial (including studies investigating LUM and/or IVA) other than Study 115B.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (17):
  - Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann & Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Respiratory and Critical Care Specialists, P.A., Children's Hospitals and Clinics of Minn, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - The Lung & Cystic Fibrosis Center at Women's & Children's Hospital of Buffalo, Buffalo, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center/Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Children's Hospital, Houston, Texas
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Canada (3):
  - British Columbia's Children's Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Centre, Glen Site, Montreal Children's Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Hoppe JE, Chilvers M, Ratjen F, McNamara JJ, Owen CA, Tian S, Zahigian R, Cornell AG, McColley SA. Long-term safety of lumacaftor-ivacaftor in children aged 2-5 years with cystic fibrosis homozygous for the F508del-CFTR mutation: a multicentre, phase 3, open-label, extension study. Lancet Respir Med. 2021 Sep;9(9):977-988. doi: 10.1016/S2213-2600(21)00069-2. Epub 2021 May 6. PMID 33965000

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was planned to have 2 cohorts: Treatment Cohort and Observational Cohort. Only the Treatment Cohort is presented in results as there were no participants enrolled in the Observational Cohort.
Pre-assignment Details: This study was conducted in participants with cystic fibrosis (CF) aged 2 years and older who participated in parent study VX15-809-115 Part B (NCT02797132).
Period: Overall Study
Arm/Group | LUM/IVA
Started | 57
Study 115B FAS (Participants enrolled and exposed to any amount of study drug in parent study VX15-809-115.) | 60
Study 116 FAS (Participants enrolled and exposed to any amount of study drug in current study VX16-809-116.) | 57
Study 116 LCI Substudy Set | 31
Completed | 47
Not Completed | 10
Not completed — Adverse Event | 2
Not completed — Withdrawal of consent (not due to AE) | 1
Not completed — Physician Decision | 2
Not completed — Commercial drug is available | 5

BASELINE CHARACTERISTICS:
Arm/Group | LUM/IVA
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: months] | 43.2 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 54
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 56
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety as Assessed by Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 98
Population: Study 116 safety set included all participants dosed in study 115B who were exposed to any amount of study drug in current study 116 treatment cohort.
Measure: Number; unit: participants
Arm/Group | LUM/IVA
Number analyzed (Participants) | 57
participants
  Participants with AEs | 56
  Participants with SAEs | 15

2. Secondary Outcome: Absolute Change in Sweat Chloride
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Parent Study 115B Baseline at Week 96
Population: Study 116 Full Analysis Set (FAS) included all participants who were enrolled and exposed to any amount of study drug in current study 116.
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | LUM/IVA
Number analyzed (Participants) | 57
millimole per liter (mmol/L) | -29.6 (12.7)

3. Secondary Outcome: Absolute Change in Body Mass Index (BMI)
Description: BMI was defined as weight in kilogram (kg) divided by height in square meter (m^2).
Time Frame: From Parent Study 115B Baseline at Week 96
Population: Study 116 FAS.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | LUM/IVA
Number analyzed (Participants) | 57
kg/m^2 | 0.30 (1.21)

4. Secondary Outcome: Absolute Change in BMI-for-age Z-score
Description: BMI was defined as weight in kilograms divided by height in m^2. z-score is a statistical measure to describe whether a mean was above or below the standard. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean.
Time Frame: From Parent Study 115B Baseline at Week 96
Population: Study 116 FAS.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | LUM/IVA
Number analyzed (Participants) | 57
z-score | 0.27 (0.73)

5. Secondary Outcome: Absolute Change in Weight
Time Frame: From Parent Study 115B Baseline at Week 96
Population: Study 116 FAS.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | LUM/IVA
Number analyzed (Participants) | 57
kg | 6.0 (2.0)

6. Secondary Outcome: Absolute Change in Weight-for-age Z-score
Description: Z-score is a statistical measure to describe whether a mean was above or below the standard. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean.
Time Frame: From Parent Study 115B Baseline at Week 96
Population: Study 116 FAS.
Measure: Mean (Standard Error); unit: z-score
Arm/Group | LUM/IVA
Number analyzed (Participants) | 57
z-score | 0.23 (0.56)

7. Secondary Outcome: Absolute Change From Baseline in Stature (Height)
Time Frame: From Parent Study 115B Baseline at Week 96
Population: Study 116 FAS.
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | LUM/IVA
Number analyzed (Participants) | 57
centimeter | 16.1 (2.3)

8. Secondary Outcome: Absolute Change in Stature-for-age Z-score
Description: as for outcome 6
Time Frame: From Parent Study 115B Baseline at Week 96
Population: Study 116 FAS.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | LUM/IVA
Number analyzed (Participants) | 57
z-score | 0.07 (0.39)

9. Secondary Outcome: Time-to-first Pulmonary Exacerbation
Description: Pulmonary exacerbation was defined as new or changed treatment with oral, inhaled, or intravenous antibiotics and fulfillment of pre-specified protocol-defined criteria.
Time Frame: From Parent Study 115B Baseline through Week 96
Population: Study 115B FAS included all participants who were enrolled and exposed to any amount of study drug in parent study 115B
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | LUM/IVA
Number analyzed (Participants) | 60
days | 600.0 [98.0 to NA] — Upper limit of inter-quartile range could not be estimated because less than 75% of participants had events.

10. Secondary Outcome: Number of Pulmonary Exacerbations (PEx)
Description: as for outcome 9
Time Frame: From Parent Study 115B Baseline through Week 96
Population: Study 115B FAS.
Measure: Number; unit: pulmonary exacerbation events
Arm/Group | LUM/IVA
Number analyzed (Participants) | 60
pulmonary exacerbation events | 82

11. Secondary Outcome: Number of Cystic Fibrosis (CF) Related Hospitalizations
Time Frame: From Parent Study 115B Baseline through Week 96
Population: Study 115B FAS.
Measure: Number; unit: hospitalizations
Arm/Group | LUM/IVA
Number analyzed (Participants) | 60
hospitalizations | 28

12. Secondary Outcome: Absolute Change in Fecal Elastase-1 (FE-1) Levels
Time Frame: From Parent Study 115B Baseline at Week 96
Population: Study 116 FAS.
Measure: Mean (Standard Deviation); unit: microgram per gram (mcg/g)
Arm/Group | LUM/IVA
Number analyzed (Participants) | 57
microgram per gram (mcg/g) | 132.6 (174.2)

13. Secondary Outcome: Absolute Change in Immunoreactive Trypsinogen (IRT) Serum Levels
Time Frame: From Parent Study 115B Baseline at Week 96
Population: Study 116 FAS.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | LUM/IVA
Number analyzed (Participants) | 57
nanogram per milliliter (ng/mL) | -108.5 (306.6)

14. Secondary Outcome: Number of Participants With Microbiology Culture Status (Positive or Negative)
Description: Following microbial tests were performed: Burkholderia, Methicillin Resistant Staphylococcus Aureus (MRSA), Methicillin Susceptible Staphylococcus Aureus (MSSA), Pseudomonas Aeruginosa Mucoid (P. Aeruginosa Mucoid), P. Aeruginosa Non-Mucoid, P. Aeruginosa Small Colony Variant and Stenotrophomonas Maltophilia.
Time Frame: Week 96
Population: Study 116 FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome at Week 96.
Measure: Number; unit: participants
Arm/Group | LUM/IVA
Number analyzed (Participants) | 46
participants
  Burkholderia (Positive) | 0
  Burkholderia (Negative) | 46
  MRSA (Positive) | 4
  MRSA (Negative) | 42
  MSSA (Positive) | 15
  MSSA (Negative) | 31
  P. Aeruginosa Mucoid (Positive) | 0
  P. Aeruginosa Mucoid (Negative) | 46
  P. Aeruginosa Non-Mucoid (Positive) | 1
  P. Aeruginosa Non-Mucoid (Negative) | 45
  P. Aeruginosa Small Colony Variant (Positive) | 0
  P. Aeruginosa Small Colony Variant (Negative) | 46
  Stenotrophomonas Maltophilia (Positive) | 2
  Stenotrophomonas Maltophilia (Negative) | 44

15. Secondary Outcome: Absolute Change in Lung Clearance Index (LCI) 2.5
Description: LCI 2.5 represents the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/40th of its starting value.
Time Frame: From Parent Study 115B Baseline at Week 96
Population: Study 116 LCI substudy set included all participants who signed the informed consent/assent to the optional LCI substudy and were enrolled and exposed to any amount of study drug in current study 116.
Measure: Mean (Standard Deviation); unit: lung clearance index
Arm/Group | LUM/IVA
Number analyzed (Participants) | 31
lung clearance index | -0.20 (1.55)

16. Secondary Outcome: Absolute Change in Lung Clearance Index (LCI) 5.0
Description: LCI 5.0 represents the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/20th of its starting value.
Time Frame: From Parent Study 115B Baseline at Week 96
Population: Study 116 LCI substudy set.
Measure: Mean (Standard Deviation); unit: lung clearance index
Arm/Group | LUM/IVA
Number analyzed (Participants) | 31
lung clearance index | 0.11 (0.65)

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 98
Arm/Group | LUM/IVA
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 15/57
Other Adverse Events (participants affected / at risk) | 55/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LUM/IVA (N=57)
Constipation (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 1
Chronic sinusitis (Infections and infestations) | 1
Gastritis viral (Infections and infestations) | 1
Gastroenteritis adenovirus (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 6
Pneumonia (Infections and infestations) | 2
Respiratory tract infection viral (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Weight gain poor (Metabolism and nutrition disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LUM/IVA (N=57)
Ear pain (Ear and labyrinth disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 17
Fatigue (General disorders) | 5
Pyrexia (General disorders) | 23
Vessel puncture site pain (General disorders) | 4
Conjunctivitis (Infections and infestations) | 4
Ear infection (Infections and infestations) | 12
Hand-foot-and-mouth disease (Infections and infestations) | 3
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 10
Influenza (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 8
Otitis media (Infections and infestations) | 7
Pharyngitis streptococcal (Infections and infestations) | 6
Pneumonia (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 12
Upper respiratory tract infection (Infections and infestations) | 13
Viral upper respiratory tract infection (Infections and infestations) | 4
Alanine aminotransferase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 5
Forced expiratory volume decreased (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 4
Pseudomonas test positive (Investigations) | 9
Staphylococcus test positive (Investigations) | 12
Decreased appetite (Metabolism and nutrition disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 47
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 25
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 18
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 5
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT03125395/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT03125395/SAP_001.pdf